CLINICAL TRIAL: NCT05209360
Title: Heel Wedges and Carbon Fiber Custom Dynamic Orthoses to Control Knee Biomechanics
Acronym: CDOKNEEpilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jason Wilken, Director of Collaborative Research and Development, Associate Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 202112360
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Adult ALL; Healthy
Keywords: Gait Analysis; Ankle Foot Orthosis; Carbon Fiber; Biomechanics; Knee Osteoarthritis
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants will be evaluated without a CDO (NoCDO), with a CDO and no wedge (CDO), with a CDO and a wedge placed on the medial aspect of the shoe (Medial), and with a CDO and a wedge placed on the lateral aspect of the shoe (Lateral)
Who Masked: Participant
Masking Description: Participants will be blinded to the testing conditions to the greatest extent possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Arm 1 (Experimental): Testing Order: NoCDO, CDO, Lateral, Medial
  Interventions: Device: Medial or Lateral Wedge; Device: Carbon Fiber Custom Dynamic Orthosis
- Arm 2 (Experimental): Testing Order: NoCDO, CDO, Medial, Lateral
  Interventions: Device: Medial or Lateral Wedge; Device: Carbon Fiber Custom Dynamic Orthosis
- Arm 3 (Experimental): Testing Order: NoCDO, Medial, CDO, Lateral
  Interventions: Device: Medial or Lateral Wedge; Device: Carbon Fiber Custom Dynamic Orthosis
- Arm 4 (Experimental): Testing Order: NoCDO, Medial, Lateral, CDO
  Interventions: Device: Medial or Lateral Wedge; Device: Carbon Fiber Custom Dynamic Orthosis
- Arm 5 (Experimental): Testing Order: NoCDO, Lateral, Medial, CDO
  Interventions: Device: Medial or Lateral Wedge; Device: Carbon Fiber Custom Dynamic Orthosis
- Arm 6 (Experimental): Testing Order: NoCDO, Lateral, CDO, Medial
  Interventions: Device: Medial or Lateral Wedge; Device: Carbon Fiber Custom Dynamic Orthosis

INTERVENTIONS:
Device: Medial or Lateral Wedge — A foam wedge that is placed inside the shoe under the CDO, that runs along the length of the foot. The tall side of the wedge will be placed on the medial (Medial Wedge) or lateral (Lateral Wedge) aspect of the shoe to preferentially load the medial or lateral side of the foot.
Device: Carbon Fiber Custom Dynamic Orthosis — A device that consists of a proximal cuff that wraps around the leg just below the knee, a posterior strut that runs the length of the leg, and a semi-rigid footplate that goes under the length of the foot.
  Other Names: CDO

SUMMARY:
The proposed study evaluates the effect of medial and lateral wedges and carbon fiber custom dynamic orthoses (CDOs) on lower limb forces and motion during walking. Previous work has used foam wedges of different stiffness and height placed under the heel to alter CDO alignment and alter lower limb mechanics. Medial or lateral wedges have been used by individuals with unilateral knee osteoarthritis in effort to reduce knee loading. In this study, medial and lateral wedges will be placed in participants shoes, with the tall side of the wedge placed on the medial or lateral aspect of the shoes, and participants will walk at controlled and self-selected speeds and complete physical performance measures. Participants will also walk without a CDO. The proposed study will provide evidence that can be used by physicians when treating knee osteoarthritis.

DETAILED DESCRIPTION:
The primary purpose of this line of research is to investigate the effects of combined carbon fiber custom dynamic orthosis (CDO) and medial or lateral wedge use on biomechanics during gait in effort to reduce unilateral knee compartment loading. The medial or lateral wedges are composed of foam, run the length of the foot, and will be placed so the tall side of the wedge is on the medial (Medial Wedge) or lateral (Lateral Wedge) aspect of the shoe to preferentially load the medial and lateral edges of the foot respectively. The use of medial and lateral wedges to treat unilateral knee osteoarthritis (OA) has been studied previously, generally without combined use of a foot and ankle brace such as a CDO. Previous work has demonstrated that foam wedges, of different height and stiffness, placed under the heel of a CDO affects sagittal plane gait biomechanics, including ankle plantarflexion and knee extension moments. The additional support and restriction of motion at the ankle associated with CDO use may emphasize results seen at the knee with medial or lateral wedging. Therefore, the proposed effort is designed to evaluate how different medial or lateral wedges placed under a CDO influence frontal plane knee biomechanics during level over-ground gait and physical performance during tests of agility, speed, and lower limb power. The proposed study will provide evidence that can be used by physicians when treating knee osteoarthritis.

In this research study, data will be collected from a cohort of healthy adult participants with no history of lower limb injuries or functional deficits. Participants will be evaluated using a series of study measures under each of the four conditions; without a brace (NoCDO), with a brace and no wedge (CDO), with a brace and a medial wedge placed in the shoe (Medial), and with a brace and a lateral wedge placed in the shoe (Lateral). The wedge will be placed in a medial and lateral position to determine effectiveness of combined wedging and CDO use in treating both medial and lateral knee OA. Testing will be randomized for each participant. Participants will walk on a level-ground walkway at self-selected and controlled speeds. Physical performance measures will incorporate tests of agility, speed, and lower limb power to ensure that the CDO and wedge do not negatively affect physical function. Questionnaires will be used to evaluate participants' pain and perception of comfort and smoothness for each testing condition.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 45
* Healthy without current complaint of lower extremity pain, spine pain, open wounds or active infections, or medical or neuromusculoskeletal disorders that have limited their participation in work or exercise in the last 6 months
* Able to hop without pain
* Able to perform a full squat without pain
* Ability to speak and understand English

Exclusion Criteria:

* Medical or neuromusculoskeletal disorders that have limited their participation in work or exercise in the last 6 months
* Diagnosed with a moderate or severe brain injury
* Lower extremity injury resulting in surgery or limiting function for greater than 6 weeks
* Injuries that would limit performance in this study
* Diagnosed with a physical or psychological condition that would preclude functional testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
* Uncorrected visual or hearing impairment(s)
* Require use of an assistive device
* Unhealed wounds (cuts/abrasions) that would prevent CDO use
* BMI > 35
* Pregnancy - Per participant self-report. Due to the expected small number of pregnant individuals, and resulting inability to account for its effect on resulting outcomes participants will be withdrawn from the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants completed study activities in each of the experimental conditions (NoCDO, CDO, Medial, Lateral) in a randomized order.
Groups:
- NoCDO, CDO, Lateral, Medial: Testing Order: NoCDO, CDO, Lateral, Medial
  Medial or Lateral Wedge: A foam wedge that is placed inside the shoe under the CDO, that runs along the length of the foot. The tall side of the wedge will be placed on the medial (Medial Wedge) or lateral (Lateral Wedge) aspect of the shoe to preferentially load the medial or lateral side of the foot.
  Carbon Fiber Custom Dynamic Orthosis: A device that consists of a proximal cuff that wraps around the leg just below the knee, a posterior strut that runs the length of the leg, and a semi-rigid footplate that goes under the length of the foot.
- NoCDO, CDO, Medial, Lateral: Testing Order: NoCDO, CDO, Medial, Lateral
  Medial or Lateral Wedge: A foam wedge that is placed inside the shoe under the CDO, that runs along the length of the foot. The tall side of the wedge will be placed on the medial (Medial Wedge) or lateral (Lateral Wedge) aspect of the shoe to preferentially load the medial or lateral side of the foot.
  Carbon Fiber Custom Dynamic Orthosis: A device that consists of a proximal cuff that wraps around the leg just below the knee, a posterior strut that runs the length of the leg, and a semi-rigid footplate that goes under the length of the foot.
- NoCDO, Medial, CDO, Lateral: Testing Order: NoCDO, Medial, CDO, Lateral
  Medial or Lateral Wedge: A foam wedge that is placed inside the shoe under the CDO, that runs along the length of the foot. The tall side of the wedge will be placed on the medial (Medial Wedge) or lateral (Lateral Wedge) aspect of the shoe to preferentially load the medial or lateral side of the foot.
  Carbon Fiber Custom Dynamic Orthosis: A device that consists of a proximal cuff that wraps around the leg just below the knee, a posterior strut that runs the length of the leg, and a semi-rigid footplate that goes under the length of the foot.
- NoCDO, Medial, Lateral, CDO: Testing Order: NoCDO, Medial, Lateral, CDO
  Medial or Lateral Wedge: A foam wedge that is placed inside the shoe under the CDO, that runs along the length of the foot. The tall side of the wedge will be placed on the medial (Medial Wedge) or lateral (Lateral Wedge) aspect of the shoe to preferentially load the medial or lateral side of the foot.
  Carbon Fiber Custom Dynamic Orthosis: A device that consists of a proximal cuff that wraps around the leg just below the knee, a posterior strut that runs the length of the leg, and a semi-rigid footplate that goes under the length of the foot.
- NoCDO, Lateral, Medial, CDO: Testing Order: NoCDO, Lateral, Medial, CDO
  Medial or Lateral Wedge: A foam wedge that is placed inside the shoe under the CDO, that runs along the length of the foot. The tall side of the wedge will be placed on the medial (Medial Wedge) or lateral (Lateral Wedge) aspect of the shoe to preferentially load the medial or lateral side of the foot.
  Carbon Fiber Custom Dynamic Orthosis: A device that consists of a proximal cuff that wraps around the leg just below the knee, a posterior strut that runs the length of the leg, and a semi-rigid footplate that goes under the length of the foot.
- NoCDO, Lateral, CDO, Medial: Testing Order: NoCDO, Lateral, CDO, Medial
  Medial or Lateral Wedge: A foam wedge that is placed inside the shoe under the CDO, that runs along the length of the foot. The tall side of the wedge will be placed on the medial (Medial Wedge) or lateral (Lateral Wedge) aspect of the shoe to preferentially load the medial or lateral side of the foot.
  Carbon Fiber Custom Dynamic Orthosis: A device that consists of a proximal cuff that wraps around the leg just below the knee, a posterior strut that runs the length of the leg, and a semi-rigid footplate that goes under the length of the foot.
Period: Overall Study
Arm/Group | NoCDO, CDO, Lateral, Medial | NoCDO, CDO, Medial, Lateral | NoCDO, Medial, CDO, Lateral | NoCDO, Medial, Lateral, CDO | NoCDO, Lateral, Medial, CDO | NoCDO, Lateral, CDO, Medial
Started | 5 | 3 | 3 | 5 | 2 | 2
Completed | 5 | 3 | 2 | 5 | 2 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study population consisted of healthy individuals ages 18-45 who met all of the study inclusion and none of the study exclusion criteria. All participants completed study activities in each of the testing conditions (NoCDO, CDO, Medial, Lateral) in a randomized order.
Groups:
- Total: Total of all reporting groups
Arm/Group | NoCDO, CDO, Lateral, Medial | NoCDO, CDO, Medial, Lateral | NoCDO, Medial, CDO, Lateral | NoCDO, Medial, Lateral, CDO | NoCDO, Lateral, Medial, CDO | NoCDO, Lateral, CDO, Medial | Total
Number analyzed (Participants) | 5 | 3 | 3 | 5 | 2 | 2 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Between 18 and 65 years | 4 | 2 | 3 | 5 | 2 | 2 | 18
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (4.5) | 26 (9.8) | 20.0 (1.0) | 23.4 (3.0) | 22.5 (4.9) | 34.5 (14.8) | 25.0 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 1 | 2 | 9
  Male | 3 | 2 | 1 | 4 | 1 | 0 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 4 | 2 | 2 | 5 | 2 | 2 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 3 | 3 | 4 | 2 | 2 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Knee Range of Motion
Description: Participants completed a biomechanical gait analysis session in all testing conditions (NoCDO, CDO Only, Medial, Lateral). Retro-reflective markers were placed on the participants skin and 12 infrared motion capture cameras (120Hz, Vicon Ltd., Oxford, UK) were used to evaluate the motion of the lower limb as participants walked at a controlled walking speed based on leg length. A minimum of three gait cycles were used to calculate mean(SD) values. Sagittal plane knee range of motion (degrees) was measured throughout the gait cycle.
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- NoCDO: Participants completed testing without an orthosis or wedge, wearing shoes only.
- CDO Only: Participants completed testing while wearing a CDO with no wedges.
  Carbon Fiber Custom Dynamic Orthosis (CDO): A device that consists of a proximal cuff that wraps around the leg just below the knee, a posterior strut that runs the length of the leg, and a semi-rigid footplate that goes under the length of the foot.
- Medial: Participants completed testing while wearing a CDO with a Medial wedges placed under the CDO footplate. The Medial wedge elevated the medial edge of the foot.
  Carbon Fiber Custom Dynamic Orthosis (CDO): A device that consists of a proximal cuff that wraps around the leg just below the knee, a posterior strut that runs the length of the leg, and a semi-rigid footplate that goes under the length of the foot.
- Lateral: Participants completed testing while wearing a CDO with a Lateral wedges placed under the CDO footplate. The Lateral wedge elevated the lateral edge of the foot.
  Carbon Fiber Custom Dynamic Orthosis (CDO): A device that consists of a proximal cuff that wraps around the leg just below the knee, a posterior strut that runs the length of the leg, and a semi-rigid footplate that goes under the length of the foot.
Arm/Group | NoCDO | CDO Only | Medial | Lateral
Number analyzed (Participants) | 20 | 20 | 20 | 19
degrees | 69.1 (4.7) | 67.0 (5.3) | 66.4 (4.7) | 66.1 (4.4)

2. Primary Outcome: Peak Knee Moment
Description: Participants completed a biomechanical gait analysis session in all testing conditions (NoCDO, CDO Only, Medial, Lateral). Retro-reflective markers were placed on the participants skin and 12 infrared motion capture cameras (120Hz, Vicon Ltd., Oxford, UK) and three force plates (1200Hz, AMTI Inc., Watertown, MA) were used to evaluate the motion and loading of the lower limb as participants walked at a controlled walking speed based on leg length. A minimum of three gait cycles were used to calculate mean(SD) values. Peak knee valgus moment was measured during stance phase and normalized to the participants body weight (Nm/kg).
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | NoCDO | CDO Only | Medial | Lateral
Number analyzed (Participants) | 20 | 20 | 20 | 19
Nm/kg | 0.4 (0.1) | 0.4 (0.1) | 0.5 (0.1) | 0.3 (0.1)

3. Primary Outcome: Four Square Step Test (4SST)
Description: The 4SST (s) is a standardized timed test of balance and agility. Participants start in the lower left quadrant of a Maltese cross setting on the floor and are timed as they move counterclockwise (forward, right, backward, left) and then clockwise (right, forward, left, backward) around the cross. Participants are instructed to move as quickly as they safely can.
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | NoCDO | CDO Only | Medial | Lateral
Number analyzed (Participants) | 19 | 19 | 19 | 19
seconds | 5.6 (0.9) | 5.8 (1.0) | 5.7 (1.0) | 5.8 (1.0)

4. Primary Outcome: Numerical Pain Rating Scale
Description: Pain will be assessed using a standard 11-point numerical pain rating scale (NPRS), in which 0 = no pain and 10 = worst pain imaginable.
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NoCDO | CDO Only | Medial | Lateral
Number analyzed (Participants) | 20 | 20 | 20 | 19
units on a scale | 0.0 (0.0) | 0.3 (0.7) | 0.6 (1.1) | 0.3 (0.6)

5. Primary Outcome: Modified Socket Comfort Score (Comfort)
Description: Participants were asked to rate the comfort of each braced condition (CDO Only, Medial, Lateral) on a scale from 0-10 with 0 = most uncomfortable to 10 = most comfortable.
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDO Only | Medial | Lateral
Number analyzed (Participants) | 20 | 20 | 19
units on a scale | 7.4 (2.2) | 6.7 (2.6) | 6.7 (2.6)

6. Primary Outcome: Modified Socket Comfort Score (Smoothness)
Description: Participants were asked to rate the smoothness of each braced condition (CDO Only, Medial, Lateral) on a scale from 0-10 with 0 = most smooth to 10 = least smooth.
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDO Only | Medial | Lateral
Number analyzed (Participants) | 20 | 20 | 19
units on a scale | 6.9 (1.9) | 6.7 (2.1) | 6.8 (2.4)

7. Secondary Outcome: Ankle Range of Motion
Description: Participants completed a biomechanical gait analysis session in all testing conditions (NoCDO, CDO Only, Medial, Lateral). Retro-reflective markers were placed on the participants skin and 12 infrared motion capture cameras (120Hz, Vicon Ltd., Oxford, UK) were used to evaluate the motion of the lower limb as participants walked at a controlled walking speed based on leg length. A minimum of three gait cycles were used to calculate mean(SD) values. Sagittal plane ankle range of motion (degrees) was measured throughout the gait cycle.
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | NoCDO | CDO Only | Medial | Lateral
Number analyzed (Participants) | 20 | 20 | 20 | 19
degrees | 32.9 (4.0) | 14.0 (3.1) | 14.9 (3.0) | 15.0 (3.2)

8. Secondary Outcome: Peak Ankle Moment
Description: Participants completed a biomechanical gait analysis session in all testing conditions (NoCDO, CDO Only, Medial, Lateral). Retro-reflective markers were placed on the participants skin and 12 infrared motion capture cameras (120Hz, Vicon Ltd., Oxford, UK) and three force plates (1200Hz, AMTI Inc., Watertown, MA) were used to evaluate the motion and loading of the lower limb as participants walked at a controlled walking speed based on leg length. A minimum of three gait cycles were used to calculate mean(SD) values. Peak ankle plantarflexor moment was measured during stance phase and normalized to the participants body weight (Nm/kg).
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | NoCDO | CDO Only | Medial | Lateral
Number analyzed (Participants) | 20 | 20 | 20 | 19
Nm/kg | 1.4 (0.1) | 1.4 (0.1) | 1.4 (0.1) | 1.4 (0.1)

9. Secondary Outcome: Peak Ankle Power
Description: Participants completed a biomechanical gait analysis session in all testing conditions (NoCDO, CDO Only, Medial, Lateral). Retro-reflective markers were placed on the participants skin and 12 infrared motion capture cameras (120Hz, Vicon Ltd., Oxford, UK) and three force plates (1200Hz, AMTI Inc., Watertown, MA) were used to evaluate the motion and loading of the lower limb as participants walked at a controlled walking speed based on leg length. A minimum of three gait cycles were used to calculate mean(SD) values. Peak ankle push-off power was measured during stance phase and normalized to the participants body weight (W/kg).
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | NoCDO | CDO Only | Medial | Lateral
Number analyzed (Participants) | 20 | 20 | 20 | 19
W/kg | 3.2 (0.5) | 1.4 (0.3) | 1.4 (0.3) | 1.5 (0.3)

10. Secondary Outcome: Sit to Stand 5 Times (STS5)
Description: STS5 (s) is a well-established timed measure of lower limb muscle strength and power. Participants are timed as they stand up and sit down 5 times as fast as possible.
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | NoCDO | CDO Only | Medial | Lateral
Number analyzed (Participants) | 19 | 19 | 19 | 19
seconds | 6.4 (1.1) | 7.4 (1.5) | 7.4 (1.6) | 7.2 (1.7)

11. Other Pre Specified Outcome: Semi-Structured Interview
Description: Semi-structured interviews will also be used to fully capture the patients' perspectives, experience, and opinions associated with the testing conditions they experienced as part of the study.
Time Frame: Baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Center of Pressure Velocity Timing
Description: Timing of peak center of pressure velocity (percent stance) during gait.
Time Frame: Baseline
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Center of Pressure Velocity Magnitude
Description: Magnitude of peak center of pressure velocity (m/s) during gait.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study participants were monitored/assessed for adverse advents throughout the duration of the study visit, up to 4 hours. Participants were also instructed to call or email the research team if any adverse events related to the study occurred after completion of the study visit, up to 6 months.
Description: [Not Specified]
Arm/Group | NoCDO | CDO Only | Medial | Lateral
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20 | 1/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NoCDO (N=20) | CDO Only (N=20) | Medial (N=20) | Lateral (N=20)
Discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — One participant found the CDO uncomfortable during walking and only completed testing in three of the four conditions. The participant indicated that the discomfort stopped after removing the CDO and that they had no lasting negative effects.

LIMITATIONS AND CAVEATS:
[Not Specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT05209360/Prot_SAP_000.pdf